CLINICAL TRIAL: NCT04578639
Title: Ocrelizumab VErsus Rituximab Off-Label at the Onset of Relapsing
Brief Title: Ocrelizumab VErsus Rituximab Off-Label at the Onset of Relapsing MS Disease
Acronym: OVERLORD-MS
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: University Hospital, Akershus (Other); Oslo University Hospital (Other); Helse Stavanger HF (Other Government); St. Olavs Hospital (Other); University Hospital of North Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020-001205-23
Record Dates: First submitted 2020-09-22; First posted 2020-10-08 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Relapsing Remitting Multiple Sclerosis
Keywords: RRMS; MS
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Rituximab; ocrelizumab

STUDY DESIGN:
Intervention Model Description: A prospective randomized double blinded multicenter non-inferiority study designed to establish non-inferiority of the study treatment rituximab compared with the comparator ocrelizumab for consecutively included patients (male or female) with active relapsing-remitting multiple sclerosis aged 18-60 years.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The investigators as well as the study participants, are blinded to the treatment allocation status. To assure this double-blinding, a dedicated "treating nurse" will be appointed at each study centre. Information about randomization (treatment arm) will be given directly through electronic communication (automatic generated email) from Viedoc™ to the treating nurse as soon as the randomization procedure has been performed. Only the treating nurse will have access to information concerning which treatment arm the patient is allocated to.
  The treating nurse will order the medicine from the pharmacy and perform the dilution in NaCl (in an infusion bag).
  An evaluating nurse and evaluating neurologist (blinded to study drug) will perform the clinical evaluation of the patient while the patient receives the medication and as part of registration of study information. The evaluating neurologist and evaluating nurse will not be able to access the randomization procedure in Viedoc™.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rituximab (Experimental): Rituximab will be given as infusion at week 0, week 26, week 52, week 78, and week 104 unless there is a reason for schedule modifications (see Section 6.3). Each infusion is given over approximately 4 hours and follow local guidelines for infusion. Initial dose; 1000 mg Subsequent doses; 500 mg
  Interventions: Drug: Rituximab
- Ocrelizumab (Active Comparator): Ocrelizumab will be given as infusion at week 0, week 26, week 52, week 78, and week 104 unless there is a reason for schedule modifications (see Section 6.3). Each infusion is given over approximately 4 hours and follow local guidelines for infusion. Initial and subsequent doses; 600 mg
  Interventions: Drug: Ocrelizumab

INTERVENTIONS:
Drug: Rituximab — A prospective randomized double blinded multicenter non-inferiority study designed to establish non-inferiority of the study treatment rituximab compared with the comparator ocrelizumab for consecutively included patients (male or female) with active relapsing-remitting multiple sclerosis aged 18-60 years. Active substance is biosimilar rituximab iv infusion and comparator is ocrelizumab (Ocrevus ®) iv infusion. Both treatments are given as infusion at month 0, month 6, month 12, month 18 and month 24. Randomization rituximab: ocrelizumab is 3:2. The primary end-point is proportion of patients with no new or enlarging T2-weighted brain MRI lesions between re-baselining at month 6 and month 24.
  Other Names: mabthera
  Arms: Rituximab
Drug: Ocrelizumab — A prospective randomized double blinded multicenter non-inferiority study designed to establish non-inferiority of the study treatment rituximab compared with the comparator ocrelizumab for consecutively included patients (male or female) with active relapsing-remitting multiple sclerosis aged 18-60 years. Active substance is biosimilar rituximab iv infusion and comparator is ocrelizumab (Ocrevus ®) iv infusion. Both treatments are given as infusion at month 0, month 6, month 12, month 18 and month 24. Randomization rituximab: ocrelizumab is 3:2. The primary end-point is proportion of patients with no new or enlarging T2-weighted brain MRI lesions between re-baselining at month 6 and month 24.
  Other Names: ocrevus
  Arms: Ocrelizumab

SUMMARY:
This is a multicenter non-inferiority study, designed to establish non-inferiority of the study treatment rituximab compared with the comparator ocrelizumab for consecutively included patients (male or female) with active relapsing-remitting multiple sclerosis aged 18-60 years.

DETAILED DESCRIPTION:
The objective of the study is to demonstrate if rituximab is non-inferior to ocrelizumab with regards to efficacy and safety in treatment naïve RRMS patients, diagnosed within the last 12 months.

To test this hypothesis, the investigators aim to perform a 30-months (24 + 6 months) prospective randomized double blinded multicenter non-inferiority study to compare rituximab to ocrelizumab in RRMS.

MS disease activity as measured by brain MRI is more sensitive as compared to clinical disease activity as measured by number of relapses or disability progression. New or enlarging MRI T2 lesions is regarded an acceptable marker of disease activity, and is routinely used in clinical practice by annual examinations (Thompson, Baranzini et al. 2018) (Thompson, Banwell et al. 2018). The investigators will therefore use the proportion of patients with no new or enlarging T2-weighted brain MRI lesions from month 6 to month 24 as the primary endpoint of this study.

Secondary objectives are included to further evaluate potential the difference or similarities in effectiveness between the treatments (disability progression, relapse rate, T25FW, 9-HPT, SDMT), to evaluate the difference in safety issues (most notably hematological complications, infections, malignancies, infusion reactions and other serious adverse events) and to evaluate the difference in patient reported outcomes by evaluation of working status, fatigue, anxiety and depressive symptoms, quality of life and treatment satisfaction (EQ-5D, MSIS-29, FSMC, and SDMT). The exploratory outcomes are included to evaluate specific blood samples and plasma biomarkers for treatment response (sNFL and CD19+ cell counts) and side effects (hypogammaglobulinemia and neutropenia) of the two treatments, differences in vaccination status (pneumococcus and/or influenza) and to determine the predictive value of BICAMS for the individual patient.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients, treatment naïve, and aged between 18 and 60 years included
2. Women of childbearing potential1 (WOCBP) able and willing to use highly effective methods of birth control2 per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly for the duration of the study OR until 3 months after last dose administered.
3. A diagnosis of RRMS according to the 2017 revised diagnostic criteria of McDonald (Thompson, Banwell et al. 2018) within the last 12 months.
4. Disease activity defined as ≥ 1 relapse3 or ≥ 1 new MRI lesion during the last 12 months
5. EDSS score ≤ 4.0
6. Absence of comorbidity or drug abuse that preclude study participation
7. Able to complete treatment or follow-up visits in the study (e.g. no contraindications for MRI or plans of moving)
8. Able to understand written and spoken Norwegian or English
9. Capable of giving signed informed consent as described in Appendix 1.2 which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

1. Known hypersensitivity or other known side effects for any of the study medications, including co-medications such as high glucocorticosteroids
2. A diagnosis of primary progressive MS according to the revised diagnostic criteria of McDonald (Thompson, Banwell et al. 2018)
3. A disease course of secondary progressive MS (Lublin, Reingold et al. 2014)
4. Any ongoing infection, including tuberculosis, hepatitis virus or HIV, as well as hepatitis B surface antigen positivity and/or hepatitis C PCR positivity verified at screening visit.
5. Prior or current psychiatric illness, mental deficiency or cognitive dysfunction influencing the patient ability to make an informed consent or comply with the treatment and follow-up phases of this protocol.
6. Cardiac insufficiency, cardiomyopathy, significant cardiac dysrhythmia, unstable or advanced ischemic heart disease (NYHA III or IV)
7. Active malignancy or prior history of malignancy except localized basal cell, squamous skin cancer or carcinoma in situ of the cervix.
8. WBC < 1.5 x 109/L if not caused by a reversible effect of documented ongoing medication. If WBC < 1.5 x 109/L is caused by a reversible effect of documented ongoing medication the WBC count must be > 1,5 x 109/L before start of study treatment.
9. Platelet (thrombocyte) count < 100 x 109/L
10. ALAT and/or ASAT more than 2 times the upper normal reference limit (ULN)
11. Serum creatinine > 200 µmol/L
12. Serum bilirubin > ULN
13. Pregnancy or lactating female patients
14. Any disease that can influence the patient safety and compliance, or the evaluation of disability
15. History of serious or life-threatening infusion reaction to ocrelizumab or rituximab, if previously treated with these medications for other diseases than MS
16. Previous use of MS-therapies such as natalizumab, fingolimod, interferons, glatiramer acetate, dimethyl fumarate, teriflunomide, cladribine, rituximab, alemtuzumab, ocrelizumab, hematopoietic stem cell therapy (HSCT) or other immunosuppression therapies with long lasting effects, or any other disease modifying therapy (DMT) for MS. If any of these medications have been used against other diseases than MS, patients can be included if the medications have not been used the previous year before enrollment.
17. Currently enrolled in another investigational device or drug study, or less than 30 days since ending another investigational device or drug study (s), or receiving other investigational treatment(s). Patients participating in a purely observational trial will not be excluded.
18. Presence of metallic objects implanted in the body, or allergy to MRI contrast that would preclude the ability of the patient to safely have MRI exams
19. Current alcohol or drug dependencies

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 214 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2025-08-14 (Estimated); Study Completion 2025-09-14 (Estimated)

PRIMARY OUTCOMES:
Proportion without new MRI activity | From month 6 (re-baseline) to month 24
  Proportion of patients with no new or enlarging T2-weighted brain MRI lesions

SECONDARY OUTCOMES:
Proportion of patients with 6-months confirmed disability progression (6M-CDP) | From baseline to month 24
  Proportion of patients with 6-months confirmed disability progression (6M-CDP) as measured by the Expanded disability status scale (EDSS) (Kurtzke 1983) from baseline to month 24. CDP-EDSS defined as an increase of one point in the EDSS score confirmed after 6 months, with an absence of relapse at the time of assessment.
Proportion of patients with 6-months confirmed disability improvement (6M-CDI) | From baseline to month 24
  Proportion of patients with 6-months confirmed disability improvement (6M-CDI) as measured by the Expanded disability status scale (EDSS) (Kurtzke 1983) from baseline to month 24. CDI-EDSS is defined as a decrease of one point in the EDSS score, confirmed after 6 months, with an absence of relapse at the time of assessment.
Annual relapse rate | From baseline to month 24
  The annual relapse rate from baseline to month 24
Proportion of patients without relapses | From baseline to month 24
  Proportion of patients without relapses from baseline to month 24
Proportion of patients with 6M-CDP in T25FW | From baseline to month 24
  Proportion of patients with 6M-CDP in T25FW (Cutter, Baier et al. 1999) from baseline to month 24. 6M-CDP in T25FW is defined as patients experiencing an increase of ≥20% from baseline which is confirmed after 6 months (Bosma, Kragt et al. 2010, Motl, Cohen et al. 2017).
Proportion of patients with 6M-CDP in 9-HPT | From baseline to month 24
  Proportion of patients with 6M-CDP in 9-HPT (Cutter, Baier et al. 1999) 8.2.6) from baseline to month 24. 6M-CDP in 9HPT is defined as patients experiencing an increase of ≥20% from baseline which is confirmed after 6 months (Bosma, Kragt et al. 2010, Feys, Lamers et al. 2017).
Proportion of patients with 6M-CDP in SDMT | From baseline to month 24
  Proportion of patients with 6M-CDP in SDMT from baseline to month 24. SDMT is defined as patients experiencing a reduction of 15% from baseline which is confirmed after 6 months (Strober, DeLuca et al. 2019, Marstrand, Osterberg et al. 2020)
Proportion of patients with no new or enlarging T2-weighted brain MRI lesions | From baseline to month 6, and from baseline to month 24
  Proportion of patients with no new or enlarging T2-weighted brain MRI lesions from baseline to month 6, and from baseline to month 24
Proportion of patients without new gadolinium enhancing T1-weighted brain MRI lesions | At month 6, month 12 and month 24
  Proportion of patients without new gadolinium enhancing T1-weighted brain MRI lesions at month 6, month 12 and month 24
Change in brain volumes | From baseline to month 24 and from month 6 to month 24
  Change in brain volumes from baseline to month 24 and from month 6 to month 24
Frequency of SAE/SAR and AESI during 24 months of treatment | From baseline to month 24
  Overall safety during 24 months of treatment
The frequency of immediate and delayed infusion reactions | From baseline to month 24
  The frequency of immediate and delayed infusion reactions during 24 months of treatment
Frequency of infections | From baseline to month 24
  The frequency of infections during 24 months of treatment
The frequency any malignancies | From baseline to month 24
  The frequency any malignancies during 24 months of treatment
Change in the quality of life (MSIS-29) | From baseline to month 24
  The Multiple Sclerosis Impact Scale (MSIS-29) is a 29-item self-report measure comprising 20 items associated with a physical scale and 9 items associated with a psychological scale, also translated and validated in Norwegian.
  Patients are asked about the impact of MS on day-to-day life in the last 2 weeks. All items have 5 response options from 1 (not at all) to 5 (extremely). Each of the 2 scales are scored by adding up the responses across items, then converting to a 0 to 100 scale, where 100 indicates greater impact of disease on daily function (worse health).
Change in Health related Anxiety and Depression as measured by HADS | From baseline to month 24
  The Hospital Anxiety and Depression Scale (HADS) is a questionnaire developed to screen anxiety and depression among patients in hospital settings. It consists of two subscales, one measuring anxiety, with seven items, and another measuring depression, with seven items. The two subscales are scored separately. The scale has been validated for use among MS patients as a screening instrument for symptoms of psychological distress. Higher scores indicate higher levels of anxiety and depression.
Change in the fatigue (FSMC) | From baseline to month 24
  The Fatigue scale for motor and cognitive functions (FSMC) is a method for evaluating fatigue in multiple sclerosis and other neurological conditions. The FSMC was developed and validated on a large sample of MS patients and healthy controls and includes subscales for both physical (motor) and mental (cognitive) aspects of fatigue. It was tested against 2 other validated fatigue scales (Fatigue Severity Scale and Modified Fatigue Impact Scale), and found to have better sensitivity and specificity than either of these instruments (Penner, Raselli et al. 2009). The FSMC has also undergone linguistic validation in over 20 languages, including Norwegian.
Change in EQ-5D score | From baseline to month 24
  The EQ-5D-5L self-report questionnaire essentially consists of 2 pages comprising:
  * The descriptive system (five dimensions of health; namely mobility, self-care, usual activities, pain/discomfort, anxiety/depression). Each dimension comprises three levels (no problems, some/moderate problems/extreme problems).
  * The EQ-VAS (visual analogue scale) which records the patient's self-rated health status on a vertical graduated (0 - 100) VAS.
Change in employment status | From baseline to month 24
  Patients will be asked about employment status at each visit (according to the following criteria: employed, unemployed, part-time employed, disability pension).
The frequency of anti-drug-antibodies | From baseline to month 24
  The frequency of anti-drug-antibodies during 24 months of treatment

OTHER OUTCOMES:
Proportion of patients with hypogammaglobinemia | From baseline to month 24
  The proportion of patients with hypogammaglobinemia during 24 months of treatment
The proportion of patients with neutropenia | From baseline to month 24
  The proportion of patients with neutropenia during 24 months of treatment
Level and duration of B cell depletion | From baseline to month 24
  The level and duration of B cell depletion during 24 months of treatment
Level of CD27+ depletion | From baseline to month 24
  The level of CD27+ B memory cell depletion during 24 months of treatment
Change in serum levels of neurofilament (Nfl) | From baseline to month 24
  Change in serum levels of neurofilament (Nfl) during 24 months of treatment
Influence of different FcR genotypes | From baseline to month 24
  The influence of different FcR genotypes on B-cell depletion during 24 months of treatment
Influence of serum levels of vitamin D | From baseline to month 24
  The influence of serum levels of vitamin D on efficacy during 24 months of treatment
Change in cognition as measured by BICAMS | From baseline to month 24
  The BICAMS is a brief cognitive assessment that can be used also in study sites with staff members with no neuropsychological training (Walker, Osman et al. 2016) The tests address specific cognitive deficits that are common in MS patients, and the scales were chosen also for their psychometric qualities (reliability, validity and sensitivity) (Langdon, Amato et al. 2012). Tests must be administered during daytime, in a standardized manner, and in a quiet room. The order of tests will be fixed: the Symbol Digit Modalities Test (SDMT), Brief Visuospatial Memory Test-Revised (BVMT-R), and California Verbal Learning Test-II (CVLT-II). BICAMS has been validated for use in Norwegian MS-patients
Vaccination response | From baseline to month 24
  Vaccination response as measured by specific pneumococcus and/or influenza antibody titres in vaccinated patients during 24 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kjell-Morten Myhr, MD, Study Director — Haukeland University Hospital; Øivind Torkildsen, MD, Principal Investigator — Haukeland University Hospital
Locations (12):
- Norway (11):
  - Haukeland University Hospital, Bergen
  - Nordlandsykehuset HF, Bodø
  - Vestre Viken sykehus, Drammen
  - Sørlandet Sykehus, Kristiansand
  - Molde sjukehus, Molde
  - Sykehuset Namsos, Namsos
  - Oslo University Hospital HF, Oslo
  - Akershus University Hospital, Oslo
  - Sykehuset Telemark, Skien
  - Stavanger University Hospital HF, Stavanger
  - University Hospital North Norway, Tromsø
- Karolinska Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No